CLINICAL TRIAL: NCT05393999
Title: The SABRE Trial: A Single-arm Prospective Study Measuring Safety, Tolerability and Pharmacokinetics of Two SARS-CoV-2 Neutralising Antibodies (C135-LS and C144-LS) Amongst High-risk Special Populations of Vaccine Non-responders.
Brief Title: SABRE: A Single-arm Prospective Study Measuring Safety and Tolerability of SARS-CoV-2 Neutralising Antibodies in High-risk Populations
Acronym: SABRE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The drug was found to be ineffective against Omicron, so the study was terminated and no patients were enrolled.
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Imperial College London (Other); University of Oxford (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21HH6747; 2021-003033-10 (EudraCT Number)
Record Dates: First submitted 2021-09-01; First posted 2022-05-27 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: SARS-CoV2 Infection; SARS-CoV-2 Acute Respiratory Disease; Myeloma; Leukemia; Lymphoma; Immune Thrombocytopenia; Thrombotic Thrombocytopenic Purpura (TTP)
MeSH Terms: conditions — COVID-19; Neoplasms, Plasma Cell; Leukemia; Lymphoma; Purpura, Thrombocytopenic, Idiopathic; Purpura, Thrombotic Thrombocytopenic | interventions — ogalvibart; crexavibart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BMS-986414 and BMS-986413 (Experimental): 1. Broadly neutralising antibody:BMS-986414 This long-acting antibody will be prescribed to all participants and given as one subcutaneous injection of 200 mg.
  2. Broadly neutralising antibody: BMS-986413 This long-acting antibody will be prescribed to all participants and given as one subcutaneous injection of 200 mg
  Interventions: Biological: BMS-986414; Biological: BMS-986413

INTERVENTIONS:
Biological: BMS-986414 — Broadly neutralising antibodies BMS-986414
  Other Names: C135-LS
Biological: BMS-986413 — Broadly neutralising antibodies BMS-986413
  Other Names: C144-LS

SUMMARY:
The SABRE study is a single-arm prospective study measuring safety, tolerability and pharmacokinetics of two SARS-CoV-2 neutralising antibodies (BMS-986414 and BMS-986413) amongst high-risk special populations of vaccine non-responders. The aim is to test the hypothesis that for individuals who fail to mount a measurable immune response to a routinely offered SARS-CoV-2 prophylactic vaccine or for those who are not able to receive such a vaccine (for example those receiving a bone marrow transplant or starting chemotherapy treatment), the receipt of subcutaneous injection of two long-acting neutralising antibodies BMS-986414 and BMS-986413 will confer durable high titres and subsequent immunological protection against SARS-CoV-2 infection.120 eligible participants will be enrolled and followed up for 48 weeks after the one-time dosing visit. Primary inclusion criteria are patients age 18 years and older and either 1) have received two doses of a routine NHS standard of care SARS-Cov-2 vaccine and do not have detectable serum SARS-CoV-2 anti-spike antibodies in routine NHS assays more than two weeks post-vaccination, or do not have protective levels of antibody or 2) be ineligible to receive a SARS-CoV-2 prophylactic vaccine. This could be because they need to commence immediate systemic chemotherapy or receive bone marrow and therefore the requirement to initiate profound immune suppression. Primary objectives are to determine the safety, tolerability and detectable SARS-CoV-2 antibody by specific PPD assay in serum at 12 weeks after enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old at screening;
* Able to give informed written consent including consent to long-term follow-up;
* Willing and able to comply with visit schedule and provide blood sampling;
* Have received at least two doses of a routine NHS standard of care SARS-Cov-2 vaccine and do not have detectable serum SARS-CoV-2 anti-spike antibodies in routine NHS assays > two weeks post 2nd vaccination, including:

  1. Solid organ transplant recipients;
  2. People with specific haematological diseases;
  3. People undergoing active chemotherapy, having immunotherapy or other continuing antibody or targeted therapy that affect immune system;
  4. People with cancers of the blood or bone marrow such as leukaemia, lymphoma or myeloma who are at any stage of treatment;
  5. People who have had bone marrow or stem cell transplants in the last 6 months or who are still taking immunosuppression drugs;
  6. People who are receiving long-term immune suppression therapy for ny other condition
* Be ineligible to receive a SARS-CoV-2 prophylactic vaccine for any of the following reasons:

  1. The need to commence immediate systemic chemotherapy;
  2. The need to receive a bone-marrow and therefore the requirement to initiate profound immune suppression
* Have an estimated life expectancy of > 12 weeks;
* Females capable of becoming pregnant* must agree to use hormonal contraception, intrauterine device, intrauterine hormone-releasing system, or to complete abstinence** from at least four weeks before the first antibody injection and for 20 months after the last antibody injection

  * Females capable of becoming pregnant are defined as: fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

**Complete abstinence (defined as refraining from heterosexual intercourse) must be in line with the preferred and usual lifestyle of the participant. Barrier contraception, periodic abstinence (e.g. calendar, ovulation, symptothermal, postovulation methods), withdrawal and progestogen-only oral hormonal contraception where inhibition of ovulation is not the primary mode of action are not acceptable methods of contraception.

Exclusion Criteria:

* Current SARS-CoV-2 infection confirmed by SARS-CoV-2 RT-PCR positive result from nasopharyngeal swab within the past 10 days and up to 24 hours prior to enrolment;
* Participation in any other clinical trial of an experimental agent or any non-interventional study where additional blood draws are required; participation in observational studies is permitted. Patients in survival follow up of another clinical trial of an investigational medicinal product (CTIMP) study may be considered if more than 5 half lives have passed since last CTIMP treatment and with permission of the medical monitor for the other study;
* History of anaphylaxis or severe adverse reaction to antibody injections, or hypersensitivity to neutralising antibodies or to any constituent products or excipients thereof;
* Treatment with intravenous immunoglobulin (IVIG) or other investigational treatments planned during the duration of the trial;
* Clinically significant abnormal blood test results at screening including:

  1. Moderate to severe hepatic impairment as defined by Child-Pugh classification;
  2. ALT >5 x ULN;
  3. INR >1.5
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Experience at least one Adverse Event of Interest (AEI). | Week 12
  Number and proportion of participants who experience at least one AEI. The total number of AEIs (where multiple events per individual are counted) will also be reported.
Experience at least one Serious Adverse Event (SAE). | Week 12
  Number and proportion of participants who experience at least one SAE. The total number of SAEs (where multiple events per individual are counted) will also be reported.
Antibody level of BMS-986414 in plasma/serum, measured using the PK assay. | Week 12
  This will be summarised using the mean, alongside an appropriate measure of variability, anticipated to be 95% confidence interval.
Antibody level of BMS-986413 in plasma/serum, measured using the PK assay. | Week 12
  This will be summarised using the mean, alongside an appropriate measure of variability, anticipated to be 95% confidence interval.

SECONDARY OUTCOMES:
Proportion achieving antibody levels of BMS-986414 in plasma/serum [measured using the PK assay] above the target PK threshold (2 ug/mL). | Weeks 1, 4, 8, 12, 24
  Number and unadjusted proportion with a corresponding 95% CI.
Proportion achieving antibody levels of BMS-986413 in plasma/serum [measured using the PK assay] above the target PK threshold (2 ug/mL). | Weeks 1, 4, 8, 12, 24
  Number and unadjusted proportion with a corresponding 95% CI.
Antibody levels of BMS-986414 in plasma/serum measured using the PK assay. | Weeks 1, 4, 8, 24
  Mean levels will be plotted against time point, alongside an appropriate measure of variability, anticipated to be 95% confidence interval.
Antibody levels of BMS-986413 in plasma/serum at measured using the PK assay. | Weeks 1, 4, 8, 24
  Mean levels will be plotted against time point, alongside an appropriate measure of variability, anticipated to be 95% confidence interval.
Antibody levels of BMS-986414 in plasma/serum measured by NHS assay. | Weeks 1, 4, 8 12, 18, 24, 32, 40, 48
  Mean levels will be plotted against time point, alongside an appropriate measure of variability, anticipated to be 95% confidence interval.
Antibody levels of BMS-986413 in plasma/serum measured by NHS assay | Weeks 1, 4, 8 12, 18, 24, 32, 40, 48
  Mean levels will be plotted against time point, alongside an appropriate measure of variability, anticipated to be 95% confidence interval.
Experience at least one Adverse Event of Interest (AEI) | Day 400
  Number and proportion of participants who experience at least one AEI. The total number of AEIs (where multiple events per individual are counted) will also be reported.
Experience at least one Serious Adverse Event (SAE) | Day 400
  Number and proportion of participants who experience at least one AEI. The total number of AEIs (where multiple events per individual are counted) will also be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Cook, Principal Investigator — Imperial College NHS Trust London; Andy Peniket, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Imperial College Heathcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No